CLINICAL TRIAL: NCT05283499
Title: Opioid Analgesic Reduction Study (OARS) - Pilot
Acronym: OARS-Pilot
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: University of Illinois at Chicago (Other); University of Maryland, Baltimore (Other); University of Michigan (Other); University of Rochester (Other)
Responsible Party: Principal Investigator, Cecile A. Feldman, DMD, Professor and Dean, Rutgers School of dental Medicine, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Pro2020001891
Record Dates: First submitted 2022-02-23; First posted 2022-03-17 (Actual); Results first posted 2022-07-13 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Post Operative Pain
Keywords: Opioids; Pain Management; Analgesics
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Analgesics, Opioid; Analgesics, Non-Narcotic

STUDY DESIGN:
Intervention Model Description: A double-blind stratified randomized clinical trial is being conduct on the management of post-surgical pain after extraction of impacted third mandibular molars Subjects will be randomly assigned to either the OPIOID or NON-OPIOID group.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Analgesic is formulate in capsules. Both OPIOID and NON-OPIOID analgesic formulas are packaged in the same capsules
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Opioid (Active Comparator): Combination analgesic of hydrocodone 5mg/acetaminophen350 mg
  Interventions: Drug: OPIOID
- Non-Opioid (Active Comparator): Combination analgesic of ibuprofen 400mgacademinophen 350mg
  Interventions: Drug: NON-OPIOID

INTERVENTIONS:
Drug: OPIOID — Analgesic assignment
  Other Names: Opioid containing analgesic
  Arms: Opioid
Drug: NON-OPIOID — Analgesic assignment
  Other Names: Non-opioid contains analgesic
  Arms: Non-Opioid

SUMMARY:
The purpose of this study is to test protocols being developed for the conduct of a large sale multi-site clinical trial which will compare opioids to non-opioids for managing post-surgical impacted 3rd molar extraction pain.

DETAILED DESCRIPTION:
A double-blind stratified randomized clinical trial is being conduct on the management of post-surgical pain after extraction of impacted third mandibular molars Subjects will be randomly assigned to either the OPIOID or NON-OPIOID group.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and non-pregnant women who are at least 18 years of age, who are able to refrain from driving or operating heavy machinery while taking the study medication will be able to participate.
* Subjects who are English speaking and are able to provide consent will be considered.
* Subjects must be in generally good health and able to take ibuprofen, paracetamol (acetaminophen), and hydrocodone.

Exclusion Criteria:

Subjects who self-report the following history will be excluded from participating:

* Individual under the age of 18
* History of gastrointestinal bleeding and/or peptic ulcer
* History of renal disease (excluding kidney stones)
* History of hepatic disease
* History of bleeding disorder
* History of respiratory depression
* Any prior respiratory effect of an opioid or other anesthetic drug that required respiratory support postoperatively
* Active or untreated asthma
* History of known allergic reaction to ibuprofen, acetaminophen, hydrocodone, and/or anesthesia
* Currently taking any of the following medications:

  * CYP3A4 inhibitor, such as macrolide antibiotics (e.g., erythromycin), azole-antifungal agents (e.g., ketoconazole), and protease inhibitors (e.g., ritonavir), which may increase plasma concentrations of hydrocodone bitartrate and acetaminophen and prolong opioid adverse reactions, and which may cause potentially fatal respiratory depression
  * CNS depressants.
* Consumes 3 or more alcoholic drinks every day and/or has a history of alcoholism
* History of drug or alcohol abuse (excludes marijuana use)
* Family history of drug or alcohol abuse in a first degree relative
* Has had one or more opioid prescription filled within the past 6 months
* Currently pregnant or lactating

Patients would also be excluded due to any additional criteria that would place the individual at increased risk or preclude the individual's full compliance with or completion of the study which includes:

* Prior participation in this study
* Inability or refusal to provide informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2020-07-06 (Actual); Primary Completion 2021-03-12 (Actual); Study Completion 2021-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janine Fredericks-Younger, DMD, Study Director — Rutgers School of Dental Medicine
Locations (5):
- United States (5):
  - University of Illinois Chicago, Chicago, Illinois
  - University of Maryland, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Rutgers University, Newark, New Jersey
  - University of Rochester, Rochester, New York

IPD SHARING:
Plan to Share IPD: Yes
Upon written request to the principle investigator data will be provided as de-identified data in csv file format.
Time Frame: Data will be available after publication of primary and secondary outcomes. Data will be available for 3 years.
Access Criteria: Requester must have a valid e-mail address.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Opioid | Non-Opioid
Started | 26 | 27
Completed | 25 | 25
Not Completed | 1 | 2
Not completed — Did not receive intervention | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Opioid | Non-Opioid | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 25 | 50
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 25
  Male | 13 | 12 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 7 | 13
  Not Hispanic or Latino | 19 | 18 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 10 | 7 | 17
  White | 3 | 11 | 14
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 5 | 2 | 7
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Pain Level
Description: Average Pain (self reported by subject) rated on numeric rating scale (0=no pain, 10=worst pain imaginable)
Time Frame: 1st day
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Opioid | Non-Opioid
Number analyzed (Participants) | 25 | 25
score on a scale | 5.67 (0.59) | 4.09 (0.59)

2. Primary Outcome: Pain Level
Description: Average Pain (self reported by subject) rated on numeric rating scale (0=no pain, 10=worst pain
Time Frame: Average for the 1st and 2nd day
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Opioid | Non-Opioid
Number analyzed (Participants) | 25 | 25
score on a scale | 5.10 (0.58) | 3.57 (0.58)

3. Primary Outcome: Pain Level
Description: Pain (self reported by subject) rated on numeric rating scale (0=no pain, 10=worst pain
Time Frame: Average for the first seven days post surgery
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Opioid | Non-Opioid
Number analyzed (Participants) | 25 | 25
score on a scale | 4.00 (0.54) | 2.74 (0.54)

4. Secondary Outcome: Sleep Quality
Description: Quality of overall sleep (self reported by subject) rated on numeric rating scale (0=best possible sleep possible, 10=worst possible sleep possible)
Time Frame: 1st night
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Opioid | Non-Opioid
Number analyzed (Participants) | 25 | 25
score on a scale | 5.45 (0.69) | 3.76 (0.70)

5. Secondary Outcome: Sleep Quality
Description: as for outcome 4
Time Frame: Average for the 1st and 2nd night
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Opioid | Non-Opioid
Number analyzed (Participants) | 25 | 25
score on a scale | 5.25 (0.64) | 3.44 (0.65)

6. Secondary Outcome: Sleep Quality
Description: as for outcome 4
Time Frame: Average for the 1st, 2nd and 3rd night
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Opioid | Non-Opioid
Number analyzed (Participants) | 25 | 25
score on a scale | 4.91 (0.63) | 3.36 (0.63)

7. Secondary Outcome: Sleep Quality
Description: as for outcome 4
Time Frame: Average for the first seven nights post surgery
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Opioid | Non-Opioid
Number analyzed (Participants) | 25 | 25
score on a scale | 4.38 (0.60) | 2.89 (0.60)

8. Secondary Outcome: Pain Interference Scale (Patient Report Outcomes Measurement Information System - PROMIS 6b )
Description: Impact of pain on subject's ability to perform normal daily functions. The sum of six questions rated on a 5 point Likert Scale (1=not at all or never, 2=a little bit or rarely, 3=somewhat or sometimes, 4=quite a bit or often and 5=very much or always)
  The six questions are: 1) how much did pain interfere with your enjoyment of life, 2) how much did pain interfere with your ability to concentrate, 3) how much did pain interfere with your day to day activities, 4) how much did pain interfere with your enjoyment of recreational activities 5) how much did pain interfere with your tasks away form and home and 6) how often did pain keep you from socializing with others?
  Minimum = 6, Maximum = 30; lower is better and higher is worse outcome
Time Frame: 1st day
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Opioid | Non-Opioid
Number analyzed (Participants) | 25 | 25
score on a scale | 17.62 (1.27) | 14.34 (1.26)

9. Secondary Outcome: Pain Interference Scale (Patient Report Outcomes Measurement Information System - PROMIS 6b )
Description: as for outcome 8
Time Frame: Average for the 1st and 2nd day
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Opioid | Non-Opioid
Number analyzed (Participants) | 25 | 25
score on a scale | 16.21 (1.18) | 12.91 (1.19)

10. Secondary Outcome: Pain Interference Scale (Patient Report Outcomes Measurement Information System - PROMIS 6b )
Description: as for outcome 8
Time Frame: Average for the 1st, 2nd and 3rd day
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Opioid | Non-Opioid
Number analyzed (Participants) | 25 | 25
score on a scale | 15.50 (1.15) | 12.19 (1.16)

11. Secondary Outcome: Pain Interference Scale (Patient Report Outcomes Measurement Information System - PROMIS 6b )
Description: as for outcome 8
Time Frame: Average for the first seven days post surgery
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Opioid | Non-Opioid
Number analyzed (Participants) | 25 | 25
score on a scale | 13.74 (1.12) | 11.01 (1.13)

12. Secondary Outcome: Overall Satisfaction
Description: Subject's rating of overall satisfaction with the analgesic provided after surgery on a 5 point Likert Scale (1=very satisfied, 2=satisfied, 3=neither satisfied or dissatisfied, 4=dissatisfied, 5=very dissatisfied)
Time Frame: Average for the first seven days post surgery
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Opioid | Non-Opioid
Number analyzed (Participants) | 25 | 25
score on a scale | 2.1 (1.4) | 1.7 (0.89)

ADVERSE EVENTS:
Time Frame: Post-operative Period -- 9 Days +/- 5 days from surgery
Description: Adverse event is defined as an event which required a unexpected office visit or visit to an emergency room and could be related to study intervention
Groups:
- OPIOID: Received hydrocodone/acetaminophen
- NON-OPIOID: Received ibuprofen/acetaminophen
Arm/Group | OPIOID | NON-OPIOID
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 1/25 | 0/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OPIOID (N=25) | NON-OPIOID (N=25)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT05283499/Prot_SAP_000.pdf
  • Informed Consent Form (2020-01-09): https://cdn.clinicaltrials.gov/large-docs/99/NCT05283499/ICF_001.pdf